CLINICAL TRIAL: NCT01093976
Title: An Open-Label Study of Dronabinol, a Cannabinoid Agonist, for Obsessive Compulsive Disorder and the Obsessive-Compulsive Spectrum Disorders Trichotillomania and Pathological Skin Picking
Brief Title: Marinol in Trichotillomania or Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0909M72088
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Trichotillomania; Obsessive Compulsive Disorder
Keywords: Skin Picking; OCD; Trichotillomania; Pathological Skin Picking
MeSH Terms: conditions — Trichotillomania; Obsessive-Compulsive Disorder; Excoriation Disorder | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dronabinol (Experimental): Dronabinol (Marinol) - 2.5mg-15mg by mouth once a day for twelve-weeks
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — 2.5mg-15mg by mouth once a day for twelve-weeks
  Other Names: MARINOL

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of dronabinol in individuals with obsessive-compulsive disorder (OCD) or the obsessive-compulsive spectrum disorders, trichotillomania (TTM) or pathological skin picking (PSP). Fifteen patients with OCD, TTM, or PSP will receive 12 weeks of open-label treatment with dronabinol. The hypothesis to be tested is that dronabinol will be effective and well tolerated in patients with these disorders. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
The study consists of twelve weeks of open-label dronabinol. All eligible study subjects will be started on open-label dronabinol 2.5mg/day for 3 weeks. The dose will be increased to 5mg/day at visit 2 (Week 3), to10mg/day at visit 3 (Week 6), and to 15mg/day at Visit 4 (Week 9) unless clinical improvement is attained at a lower dose (clinical improvement will be assessed by the investigator with respect to obsessive thoughts, urges and compulsive behaviors). Subjects will be seen every three weeks during the 12-week, open-label study. All efficacy and safety assessments will be performed at each visit. Subjects who are not compliant with their use of study medication (i.e. failing to take medication for three or more consecutive days) will be discontinued from the study.

Laboratory testing, including liver function tests, a blood chemistry panel, and urine toxicology will be completed for subjects at baseline if in the opinion of the study physician the medical history of the subject warrants such tests for their safety. All females, regardless of age, will undergo a urine pregnancy test at screening and all subjects will be required to do a urine drug screen at the screening visit to test for drugs of abuse.

At study conclusion, subjects will be given the option to continue on medication (via prescription) if covered by insurance, and will then be followed in our clinic or referred to another psychiatrist. All study subjects will be offered follow-up care with CBT and/or medication in our outpatient clinic (if covered by insurance) or be given a list of appropriate referrals in the community.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Obsessive-compulsive disorder (OCD), Trichotillomania (TTM), or Pathological Skin Picking (PSP) as the primary psychiatric diagnosis
3. (If OCD) - Subject reports ≥two failed treatments using selective serotonin reuptake inhibitors (SSRIs) for their OCD
4. Women's participation required negative results on a beta-human chorionic gonadotropin pregnancy test and stable use of a medically accepted form of contraception.
5. Signed informed consent before entry into the study.

Exclusion Criteria:

1. Unstable medical illness or clinically significant abnormalities on laboratory tests or physical examination at screening visit
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. A need for medication other than dronabinol with possible psychotropic effects
4. History of hypersensitivity to any cannabinoid or sesame oil
5. Lifetime history of bipolar disorder type I or II, dementia, or schizophrenia as determined by the Structured Clinical Interview for DSM-IV
6. Current (past 12-months) DSM-IV substance abuse or dependence
7. Positive urine drug screen at screening
8. Initiation of cognitive behavior therapy within 3 months prior to study baseline
9. Baseline score of ≥ 17 on the Hamilton Depression Rating Scale (17-item HDRS
10. Suicidality based on clinical interview
11. History of head injury or neurological disorder (such as seizures)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- Ambulatory Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Grant JE, Odlaug BL, Chamberlain SR, Kim SW. Dronabinol, a cannabinoid agonist, reduces hair pulling in trichotillomania: a pilot study. Psychopharmacology (Berl). 2011 Dec;218(3):493-502. doi: 10.1007/s00213-011-2347-8. Epub 2011 May 19. PMID 21590520
- See also: Impulse Control Disorders Clinic - University of Minnesota — http://www.impulsecontroldisorders.org/index.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dronabinol
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dronabinol
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.29 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Massachusetts General Hospital Hairpulling Scale (MGH-HPS) Total Score
Description: The MGH-HPS is a 7-item, self-report scale that rates urges to pull hair, actual amount of pulling, perceived control over behavior, and distress associated with hair pulling over the past seven days. Total possible score is a 28 indicating the highest level of severity out of a scale from 0-28.
Time Frame: Subjects were followed for their duration of participation in the study (12-weeks)
Population: Mean score reported below is the endpoint MGH-HPS score (at 12-weeks or last-observation carried forward).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol
Number analyzed (Participants) | 14
units on a scale | 8.71 (5.48)

ADVERSE EVENTS:
Arm/Group | Dronabinol
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=14)
Light-headed / dizziness (Psychiatric disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No